# Optimizing Online Purchasing of Fruits, Vegetables, and Legumes for Low-Income Families

NCT07071753

Document Date: 01/22/2026

## RESEARCH INFORMED CONSENT FORM

**STUDY TITLE:** OPT-FRESH (IRB-FY2025-10110)

INVESTIGATOR(S): Angela Trude, PhD

FUNDING SPONSOR: National Institutes of Health

## INVITATION TO BE A PART OF A RESEARCH STUDY

• You are being asked to join a research study.

- This form explains what the study is about and what you would do.
- You don't have to join. It's your choice.
- If you do join, you can stop at any time. No one will be upset.
- We will tell you if anything changes that might affect your decision to stay in the study.

## **PURPOSE OF THE STUDY**

We want to learn what helps parents or caregivers buy food for their home. This study takes place in New York City. You are being asked to join because you care for a child under 10 years old. About 360 families will be in the study. The study will last about 5 years.

#### **ELIGIBILITY TO PARTICIPATE**

You are eligible to participate in this study if you:

- are 21 or older
- buy most of the food in your home
- your family gets SNAP or has low income
- are okay with ordering groceries online
- own a smartphone
- agree to share grocery receipts
- speak English or Spanish

We will ask you a few questions to make sure you qualify.

## **DESCRIPTION OF STUDY PROCEDURES**

If you join, here's what you'll be asked to do:

# **Before the Program**:

- Take a short online survey (15–20 minutes) about your food and shopping habits
- Meet us once in your community for you and your child to:
  - Have height and weight measured
  - Use a tool called a Veggie Meter to scan your skin
- Send at least two recent grocery receipts

<u>Then:</u> You'll be randomly placed into a group. This means it is done completely by chance, like pulling a name out of a hat or flipping a coin. Neither you nor the research team can choose your group. Every family has the same chance of being placed into the groups. You may be in

only one group, or in more than one group. For example, you might only be in the group that only received rewards for produce, only in the group that only receives text messages, or in both.

# **During the Program (12 weeks):**

- You get a free Instacart Express Membership (no delivery fee for orders \$10 or more) plus:
  - A text on how to use Instacart
  - A call in the first week to help you set it up
  - A packet in the mail with simple steps
- Depending on the group you are randomized in, you may also get one or a combination of the following:
  - 1. Weekly texts to guide your grocery shopping
  - 2. A \$1 reward for every \$1 you spend on fruits, veggies, and beans (up to \$10/week)
  - 3. Meal ideas and shopping lists by text and mail
- We'll also ask you to:
  - Fill out a short survey once half-way through the program,
  - Send grocery receipts once per week

# After the Program Ends:

- Online survey
- In-person visit for you and your child
- Submit at least two grocery receipts

## 9 Months Later:

- Final online survey
- Send at least two grocery receipts
- Get your Instacart Membership reactivated

## **Optional Interview:**

- 60-minute interview by phone or Zoom
- Share your experience and feedback

# **RISKS OR DISCOMFORTS**

There are no physical risks to you or your child. Some questions may make you feel uncomfortable. You can skip any question or stop at any time. If anything upsets or harms you, please tell us.

## **BENEFITS**

Being in this study may help you and your family:

- You may get helpful or interesting information in text messages or mail.
- You will get a free Instacart Express Membership to help order groceries online.

- You may learn how to use SNAP benefits online.
- It may be easier to get healthy foods, like fruits, vegetables, and beans.

We cannot promise that you will benefit, but many families find some of these things helpful.

Your help will also teach researchers how to make it easier for families to get food in your neighborhood.

## **COMPENSATION**

- 1. **Before the program starts**: upon completion of the initial survey, in-person measures, and submission of complete grocery receipts of a household shopping, you will receive a \$20 Amazon electronic gift card within 7 days.
- 2. **During the Program**: You will receive \$5 per week during the 12-week intervention period for submitting complete grocery receipts of a household shopping (in-store or online) to the research team as Instacart Fresh Funds to apply towards service fees.
- 3. **Immediately After the Program**: When you complete the online survey, in-person measures, and submit two additional weeks of grocery receipts you will receive a \$30 Amazon electronic gift card within 7 days.
- 4. **After 9 Months from the Program**: When you complete the brief online survey <u>and</u> submit at least two itemized grocery receipts, you will receive a \$20 Amazon electronic gift card within 7 days.
- 5. **Optional individual interview**: you will receive a \$20 Amazon electronic gift card within 7 days.

If you complete all steps of the program, you may receive up to \$90 Amazon electronic gift card and \$60 Instacart Fresh Funds to apply towards service fees.

#### **VOLUNTARY PARTICIPATION**

Participating in this study is completely voluntary. You may choose not to take part in the study or to stop participating at any time, for any reason, without penalty or negative consequences.

If you withdraw from the study early you will still receive gift card payments for each completed phase but will not be eligible for future incentives.

If you withdraw or are withdrawn from the study early, then we will keep information about you that is already collected.

If we learn something new during the study that might affect your decision to stay in, we will tell you right away.

# PRIVACY & DATA CONFIDENTIALITY

We will keep your information safe. Your name won't be in reports. Only the research team and certain approved groups can see your private information.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. Researchers with this Certificate will not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, even if there is a court subpoena.

Exceptions include:

- A federal, state, or local law requires disclosure.
- Your explicit approval for the researchers to release your name or any other personally identifiable information.

## Future Use of Data

Information about you collected for this study may be shared with other researchers, used for other research studies, or placed in a data repository. These studies may be similar to this study or completely different. All information that could identify you will be removed before sharing the data or using it for other research studies. We will not ask you for additional permission before sharing the information.

In the future, the program or parts of it could also be used in ways that make money, such as being part of a business or product. If that happens, it will be treated as intellectual property (like an invention or idea that belongs to the university or researchers). You will not be paid or receive any profit from this, even if the program is used or sold in the future.

## **ACCESS TO YOUR STUDY INFORMATION**

We will give you access to the information that is collected about you in this study by requesting directly from the study team. The investigator will share information with participants if there is a concern. Participants can always access their information via study applications.

# **ALTERNATIVES TO PARTICIPATING**

You do not have to join this study. If you choose not to take part, nothing will change in the care or help you already get.

If you're still interested in learning how to get food or support for your household groceries, there may be other programs in your community that can help.

If you want, we can give you a list of local programs or resources that offer similar support.

#### CONTACT INFORMATION

You are encouraged to ask questions at any time during this study. For information about the study, contact Angela Trude at 212-988-5456, at5285@nyu.edu.

If you have questions about your rights as a research participant or if you believe you have been harmed from the research, please contact the NYU Human Research Protection Program at (212)998-4808 or ask.humansubjects@nyu.edu.

# **AGREEMENT TO PARTICIPATE**

By checking below, you are agreeing to participate in this study. Make sure you understand what the study involves before you agree. If you have questions about the study after you agree to participate, you can contact the research team using the information provided above. You may [print/keep] a copy of this form.

[] I agree to participate in this research study.